CLINICAL TRIAL: NCT05007392
Title: A Randomized, Multicenter, Double-Blind, Superiority Study of Dotinurad (4 mg) and Febuxostat (40 mg) for the Treatment of Subjects With Gout
Brief Title: A Study to Evaluate Efficacy of Dotinurad and Febuxostat for the Treatment of Participants With Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYU-981-J086-301
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Gout
Keywords: Dotinurad; Febuxostat
MeSH Terms: conditions — Gout | interventions — dotinurad; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: Dotinurad + Febuxostat Matched Placebo (Experimental): Participants will receive one dotinurad 1 mg tablet and one febuxostat 20 mg matched placebo tablet, orally, once daily on Day 1 to Day 28 (up to 4 weeks) in Treatment 1 Phase; and then one dotinurad 2 mg tablet and two febuxostat 20 mg matched placebo tablets, orally, once daily on Day 29 to Day 84 (up to 8 weeks) followed by two dotinurad 2 mg tablets and two febuxostat 20 mg matched placebo tablets, orally, once daily on Day 85 to Day 168 (up to 12 weeks) in Treatment 2 Phase (Treatment 1 Phase=4 weeks; Treatment 2 Phase=20 weeks).
  Interventions: Drug: Dotinurad; Other: Febuxostat Matched Placebo
- Drug: Febuxostat + Dotinurad Matched Placebo (Active Comparator): Participants will receive one febuxostat 20 mg tablet and one dotinurad 1 mg matched placebo tablet, orally, once daily on Day 1 to Day 28 (up to 4 weeks) in Treatment 1 Phase; and then two febuxostat 20 mg tablets and one dotinurad 2 mg matched placebo tablet, orally, once daily on Day 29 to Day 84 (up to 8 weeks) followed by two febuxostat 20 mg tablets and two dotinurad 2 mg matched placebo tablets, orally, once daily on Day 85 to Day 168 (up to 12 weeks) in Treatment 2 Phase (Treatment 1 Phase=4 weeks; Treatment 2 Phase=20 weeks).
  Interventions: Drug: Febuxostat; Other: Dotinurad Matched Placebo

INTERVENTIONS:
Drug: Dotinurad — Dotinurad oral tablets.
  Other Names: FYU-981
  Arms: Drug: Dotinurad + Febuxostat Matched Placebo
Drug: Febuxostat — Febuxostat oral tablets.
  Arms: Drug: Febuxostat + Dotinurad Matched Placebo
Other: Dotinurad Matched Placebo — Dotinurad matched placebo oral tablets.
  Arms: Drug: Febuxostat + Dotinurad Matched Placebo
Other: Febuxostat Matched Placebo — Febuxostat matched placebo oral tablets.
  Arms: Drug: Dotinurad + Febuxostat Matched Placebo

SUMMARY:
The primary purpose of the study is to confirm the efficacy of dotinurad 4 milligram (mg) to febuxostat 40 mg on the percentage of participants achieving a serum uric acid (SUA) level less than or equal to (<=) 6.0 milligrams per deciliter (mg/dL) at Week 24 in Chinese participants with gout.

ELIGIBILITY:
Inclusion Criteria:

1. Gout participant (with a history of gout attack or concurrent gouty tophi) with SUA level greater than (>) 7.0 mg/dL in the screening phase (within 14 days prior to randomization)
2. Male or female participant with age greater than or equal to (>=) 18 years at the time of informed consent
3. Provide written informed consent signed by the participant prior to entering the study or undergoing any study procedures, indicating that they understand the purpose and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

1. Has gouty arthritis that has not resolved within 14 days prior to randomization
2. Has secondary hyperuricemia
3. Comorbidities with nephrolithiasis or clinical urinary calculi (example, haematuria, back pain)
4. Evidence of clinically significant disease (example, cardiac disease: heart failure and angina unstable, respiratory, gastrointestinal, renal, or neurological disease: cerebral infarction) that in the opinion of the investigator could affect the participant's safety or interfere with the study assessments
5. Evidence of clinical significant hepatic disease: refer to Grade 2 in the "Seriousness Grading Criteria for Adverse Drug Reactions" or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 multiple (*) upper limit of normal (ULN) in the screening phase
6. Estimated glomerular filtration rate (eGFR) of less than (<) 30 milliliter per minute/1.73 square meters in the screening phase
7. Systolic blood pressure of >=180 millimetre of mercury (mmHg) or diastolic blood pressure of >=110 mmHg in the screening phase
8. Hemoglobin A1c National Glycohemoglobin Standardization Program (NGSP) value of >=8.4 percent (%) in the screening phase
9. Hypersensitivity to the study drugs (dotinurad or febuxostat) or their excipients, or all of urine alkalinizer (potassium citrate/sodium citrate hydrate compound preparations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Anzhen Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tongzhou District Luhe Hospital, Beijing, P.R.China, Beijing, Beijing Municipality
  - Foshan First People's Hospital, Foshan, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - The Seventh Affiliated Hospital of Sun Yat-sen University, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The Third Xiangya Hospital of Central South University, Changsha, Hu'nan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - First Affiliated Hospital of Inner Mongolia technological University, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Nanjing Medical University Affiliated 2nd Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital, Yanji, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Dalian Municipal Central Hospital Affiliated of Dalian Medical University, Dalian, Liaoning
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tong Ren Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai, Shanghai Municipality
  - The First People's Hospital of Yunnan Province, Kunming, Yun'nan

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 30 investigative sites in China from 21 December 2021 to 14 June 2023.
Pre-assignment Details: A total of 604 participants were screened, of which 153 were screen failure. 451 participants were enrolled and randomized and 448 received study treatment.
Groups:
- Febuxostat: Participants received febuxostat 20 milligrams (mg) tablet, orally, once daily for first 4 weeks; followed febuxostat 40 mg tablet, orally, once daily for 20 weeks. To maintain blinding, participants also received the dotinurad matching placebo up to Week 24.
- Dotinurad: Participants received dotinurad 1 mg tablet, orally, once daily for first 4 weeks; followed by dotinurad 2 mg tablet, orally, once daily for 8 weeks; further followed by dotinurad 4 mg tablet, orally, once daily for 12 weeks. To maintain blinding, participants also received the febuxostat matching placebo up to Week 24.
Period: Overall Study
Arm/Group | Febuxostat | Dotinurad
Started | 226 | 225
Safety Analysis Set (Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.) | 225 | 223
Full Analysis Set (Full Analysis Set was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement.) | 220 | 221
Completed | 197 | 195
Not Completed | 29 | 30
Not completed — Randomized but not treated | 1 | 2
Not completed — Other | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Serum uric acid (SUA) level of <=2.0 milligram per deciliter (mg/dL) for 2 consecutive visits | 0 | 1
Not completed — Use of prohibited concomitant drug | 1 | 1
Not completed — Inadequate therapeutic effect or progression of disease | 1 | 0
Not completed — Adverse Event | 10 | 6
Not completed — Participant choice | 5 | 10
Not completed — Withdrawal of consent | 5 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement.
Groups:
- Febuxostat: Participants received febuxostat 20 mg tablet, orally, once daily for first 4 weeks; followed febuxostat 40 mg tablet, orally, once daily for 20 weeks. To maintain blinding, participants also received the dotinurad matching placebo up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Febuxostat | Dotinurad | Total
Number analyzed (Participants) | 220 | 221 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (10.98) | 38.9 (11.56) | 39.1 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 215 | 218 | 433
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 220 | 221 | 441
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 220 | 221 | 441
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Uric Acid (SUA) Level <=6.0 mg/dL at Week 24 (LOCF)
Description: Percentage of participants with SUA level less than or equal to (<=) 6.0 milligrams per deciliter (mg/dL) at Week 24 was reported. In case the SUA level was missing, this data was compensated by the last observation carried forward (LOCF) method.
Time Frame: At Week 24
Population: Full Analysis Set was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 218 | 220
percentage of participants | 38.1 [31.6 to 44.5] | 73.6 [67.8 to 79.5]
Statistical Analysis 1: Comparison: Febuxostat vs Dotinurad; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; P value based on a Cochran-Mantel-Haenszel test stratified by baseline SUA level and baseline body mass index (BMI) level; Difference of percentage = 35.87, 95% CI 2-sided [27.36 to 44.37] — The difference of percentage and stratified 95 percent (%) confidence interval (CI) was based on Mantel-Haenszel method

2. Secondary Outcome: Percentage of Participants With SUA Level <=6.0 mg/dL at Week 12 (LOCF)
Description: Percentage of participants with SUA level <=6.0 mg/dL at Week 12 was reported. In case the SUA level was missing, this data was compensated by the LOCF method.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 216 | 220
percentage of participants | 50.5 [43.8 to 57.1] | 55.5 [48.9 to 62.0]
Statistical Analysis 1: Comparison: Febuxostat vs Dotinurad; Test type: Non-Inferiority — The prespecified non-inferiority margin was -10% in the analysis; Difference of percentage = 5.24, 95% CI 2-sided [-3.69 to 14.17] — The difference of percentage and stratified 95% CI was based on Mantel-Haenszel method

3. Secondary Outcome: Percentage of Participants With SUA Level <=6.0 mg/dL at Weeks 4, 8, 12, 16, 20 and 24
Description: Percentage of participants with SUA level <=6.0 mg/dL at Weeks 4, 8, 12, 16, 20 and 24 was reported. Data was reported for observed participants at specified visits.
Time Frame: At Weeks 4, 8, 12, 16, 20 and 24
Population: Full Analysis Set was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, "overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 198 | 202
percentage of participants
  Week 4: number analyzed (Participants) | 198 | 196
  Week 4 | 26.3 | 27.6
  Week 8: number analyzed (Participants) | 189 | 201
  Week 8 | 55.6 | 62.7
  Wee 12: number analyzed (Participants) | 197 | 202
  Wee 12 | 52.8 | 56.9
  Week 16: number analyzed (Participants) | 195 | 196
  Week 16 | 48.7 | 84.7
  Week 20: number analyzed (Participants) | 190 | 188
  Week 20 | 53.7 | 83.0
  Week 24: number analyzed (Participants) | 189 | 192
  Week 24 | 40.2 | 78.1

4. Secondary Outcome: Mean Percent Reduction From Baseline in SUA Level at Weeks 4, 8, 12, 16, 20 and 24
Description: Mean percent reduction from baseline in SUA level at Weeks 4, 8, 12, 16, 20 and 24 was reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change in SUA level
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 198 | 202
Percent change in SUA level
  Percent Reduction from Baseline at Week 4: number analyzed (Participants) | 198 | 196
  Percent Reduction from Baseline at Week 4 | 26.43 (13.200) | 27.43 (14.754)
  Percent Reduction from Baseline at Week 8: number analyzed (Participants) | 189 | 201
  Percent Reduction from Baseline at Week 8 | 37.06 (14.018) | 39.10 (18.931)
  Percent Reduction from Baseline at Week 12: number analyzed (Participants) | 197 | 202
  Percent Reduction from Baseline at Week 12 | 36.06 (15.383) | 38.62 (17.305)
  Percent Reduction from Baseline at Week 16: number analyzed (Participants) | 195 | 196
  Percent Reduction from Baseline at Week 16 | 35.13 (16.016) | 51.47 (18.542)
  Percent Reduction from Baseline at Week 20: number analyzed (Participants) | 190 | 188
  Percent Reduction from Baseline at Week 20 | 35.71 (15.728) | 50.22 (20.714)
  Percent Reduction from Baseline at Week 24: number analyzed (Participants) | 189 | 192
  Percent Reduction from Baseline at Week 24 | 32.28 (16.907) | 48.07 (23.243)

5. Secondary Outcome: Mean Change From Baseline in SUA Level at Weeks 4, 8, 12, 16, 20 and 24
Description: Mean change from baseline in SUA level at Weeks 4, 8, 12, 16, 20 and 24 was reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 198 | 202
mg/dL
  Change from Baseline at Week 4: number analyzed (Participants) | 198 | 196
  Change from Baseline at Week 4 | -2.60 (1.457) | -2.70 (1.508)
  Change from Baseline at Week 8: number analyzed (Participants) | 189 | 201
  Change from Baseline at Week 8 | -3.62 (1.597) | -3.80 (1.973)
  Change from Baseline at Week 12: number analyzed (Participants) | 197 | 202
  Change from Baseline at Week 12 | -3.52 (1.691) | -3.78 (1.817)
  Change from Baseline at Week 16: number analyzed (Participants) | 195 | 196
  Change from Baseline at Week 16 | -3.44 (1.731) | -5.05 (2.078)
  Change from Baseline at Week 20: number analyzed (Participants) | 190 | 188
  Change from Baseline at Week 20 | -3.52 (1.757) | -4.92 (2.201)
  Change from Baseline at Week 24: number analyzed (Participants) | 189 | 192
  Change from Baseline at Week 24 | -3.20 (1.800) | -4.71 (2.415)

6. Secondary Outcome: Mean SUA Level at Baseline, Weeks 4, 8, 12, 16, 20 and 24
Description: Mean SUA level at Baseline, Weeks 4, 8, 12, 16, 20 and 24 was reported.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20 and 24
Population: Full Analysis Set was the group of randomized participants who received at least 1 dose of study drug and had at least 1 post-dose primary efficacy measurement. Here, "number analyzed" signifies those participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Febuxostat | Dotinurad
Number analyzed (Participants) | 220 | 221
mg/dL
  Baseline | 9.65 (1.426) | 9.67 (1.451)
  Week 4: number analyzed (Participants) | 198 | 196
  Week 4 | 7.07 (1.432) | 6.93 (1.447)
  Week 8: number analyzed (Participants) | 189 | 201
  Week 8 | 6.01 (1.372) | 5.80 (1.857)
  Week 12: number analyzed (Participants) | 197 | 202
  Week 12 | 6.12 (1.546) | 5.88 (1.708)
  Week 16: number analyzed (Participants) | 195 | 196
  Week 16 | 6.24 (1.605) | 4.65 (1.776)
  Week 20: number analyzed (Participants) | 190 | 188
  Week 20 | 6.14 (1.467) | 4.76 (1.900)
  Week 24: number analyzed (Participants) | 189 | 192
  Week 24 | 6.49 (1.575) | 5.00 (2.296)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 24
Description: Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Arm/Group | Febuxostat | Dotinurad
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/223
Serious Adverse Events (participants affected / at risk) | 4/225 | 3/223
Other Adverse Events (participants affected / at risk) | 203/225 | 201/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=225) | Dotinurad (N=223)
Cataract (Eye disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat (N=225) | Dotinurad (N=223)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Monocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 3 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0
Right ventricular hypertrophy (Cardiac disorders) | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Dry eye (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 1 | 0
Xerophthalmia (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 11
Toothache (Gastrointestinal disorders) | 2 | 4
Chronic gastritis (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Gingival swelling (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal eczema (Gastrointestinal disorders) | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileal ulcer (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 11 | 7
Fatigue (General disorders) | 1 | 1
Influenza like illness (General disorders) | 4 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 18 | 24
Hepatic steatosis (Hepatobiliary disorders) | 4 | 3
Liver injury (Hepatobiliary disorders) | 4 | 3
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Gallbladder enlargement (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0
COVID-19 (Infections and infestations) | 57 | 57
Upper respiratory tract infection (Infections and infestations) | 22 | 13
Coronavirus infection (Infections and infestations) | 3 | 5
Influenza (Infections and infestations) | 2 | 4
Nasopharyngitis (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 1 | 3
Bronchitis (Infections and infestations) | 0 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 2
Abscess limb (Infections and infestations) | 0 | 1
Carbuncle (Infections and infestations) | 0 | 1
Clonorchiasis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Helicobacter infection (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Tinea cruris (Infections and infestations) | 1 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 28 | 18
SARS-CoV-2 test positive (Investigations) | 8 | 17
Alpha 1 microglobulin increased (Investigations) | 19 | 12
Blood uric acid decreased (Investigations) | 1 | 10
Gamma-glutamyltransferase increased (Investigations) | 12 | 10
Blood creatine phosphokinase increased (Investigations) | 15 | 8
Blood creatinine increased (Investigations) | 8 | 7
Low density lipoprotein increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 12 | 6
Eosinophil count increased (Investigations) | 3 | 6
High density lipoprotein decreased (Investigations) | 3 | 6
Beta 2 microglobulin urine increased (Investigations) | 7 | 5
Amylase increased (Investigations) | 2 | 4
Beta 2 microglobulin increased (Investigations) | 4 | 4
Urine osmolarity decreased (Investigations) | 5 | 4
Blood cholesterol increased (Investigations) | 2 | 3
Protein urine present (Investigations) | 2 | 3
Urinary occult blood positive (Investigations) | 3 | 3
White blood cell count decreased (Investigations) | 2 | 3
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 7 | 2
Blood bilirubin increased (Investigations) | 0 | 2
Blood glucose increased (Investigations) | 4 | 2
Blood pressure diastolic increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 2
Weight increased (Investigations) | 0 | 2
Alanine aminotransferase (Investigations) | 0 | 1
Albumin urine present (Investigations) | 0 | 1
Blood glucose (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood triglycerides (Investigations) | 0 | 1
Blood triglycerides increased (Investigations) | 3 | 1
Blood urea increased (Investigations) | 0 | 1
Bone density increased (Investigations) | 1 | 1
Coronavirus test positive (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Globulins increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 1
Monocyte count decreased (Investigations) | 0 | 1
Monocyte count increased (Investigations) | 1 | 1
Renal scan abnormal (Investigations) | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 1
Weight decreased (Investigations) | 0 | 1
White blood cells urine positive (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 0
Blood glucose abnormal (Investigations) | 2 | 0
Creatinine urine increased (Investigations) | 1 | 0
Electrocardiogram P wave abnormal (Investigations) | 1 | 0
Electrocardiogram Q waves (Investigations) | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 3 | 0
Electrocardiogram repolarisation abnormality (Investigations) | 1 | 0
Globulins decreased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Urinary occult blood (Investigations) | 2 | 0
White blood cell count increased (Investigations) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 13 | 16
Gout (Metabolism and nutrition disorders) | 13 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 4
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 78 | 97
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Dreamy state (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Cardiovascular somatic symptom disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 17 | 14
Microalbuminuria (Renal and urinary disorders) | 4 | 6
Haematuria (Renal and urinary disorders) | 4 | 5
Renal cyst (Renal and urinary disorders) | 5 | 4
Renal impairment (Renal and urinary disorders) | 4 | 3
Proteinuria (Renal and urinary disorders) | 5 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Albuminuria (Renal and urinary disorders) | 1 | 1
Renal injury (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Leukocyturia (Renal and urinary disorders) | 1 | 0
Renal milk of calcium cyst (Renal and urinary disorders) | 1 | 0
Urate nephropathy (Renal and urinary disorders) | 1 | 0
Prostatic calcification (Reproductive system and breast disorders) | 4 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 7 | 5
Phlebolith (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT05007392/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT05007392/SAP_001.pdf